CLINICAL TRIAL: NCT02301871
Title: Efficacy of Muscle Energy Technique and Deep Neck Flexors Training in Mechanical Neck Pain- A Randomized Clinical Trial
Brief Title: The Effect of Soft Tissue Mobilization in Myofascial Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, HARSHITA YADAV, Efficacy of Muscle Energy Technique and Deep Neck Flexors Training in Mechanical Neck Pain- A Randomized Clinical Trial, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N44-449
Record Dates: First submitted 2014-11-22; First posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Neck Pain
Keywords: MNP; MET; Soft tissue mobilization; DNF; Static Stretching
MeSH Terms: conditions — Neck Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional group (Active Comparator): The treatment was given for 5 days per week for 2 weeks such as MHP (Moist Heat Pack) for 20 minutes, Static Stretching exercises for upper trapezius, levator scapulae and scalene muscle which is held for 10-30 seconds- repeated 3-5 times, Cervical spine non-thrust mobilization (Grade 3) was given to each segment from C2-C7 was oscillated for 10 repetitions, followed by a 10 seconds rest between segments, Cervical spine active ROM (Range of Motion) exercises with 10 repetitions- 2-3 times a day and Postural exercises were given as home programme.
  Interventions: Procedure: Static stretching and Cervical non thrust manipulation
- DNF Group (Experimental): DNF training along with conventional treatment. In this programme, emphasis was placed on first attaining the correct craniocervical flexion action, with minimal activity of the superficial cervical flexor muscles. The craniocervical flexion action involves a specific craniocervical movement (nodding - "yes" movement) of head such that it remains in contact with the supporting surface. Once the correct action had been achieved, participants were instructed in the use of the sphygmomanometer to guide the training of the CCF muscle contraction at the various incremental levels of pressure (22 to 30 mmHg, progressively inner range positions).
  Interventions: Device: Dr. Gene's Health and Wellness
- MET Group (Experimental): MET in additional to conventional treatment. MET was applied to Upper trapezius, Levator scapulae and Scalene Following the 7-10 seconds isometric contraction and complete relaxation of all elements, the stretch is maintained for 30 seconds. The effort and the counter-pressure should be modest (20% of available strength) and painless. The process is repeated 3-5 times.
  Interventions: Procedure: Muscle Energy Technique

INTERVENTIONS:
Device: Dr. Gene's Health and Wellness — The device is used to perfom deep neck flexors muscles traning. These low load craniocervical flexion exercise are even in early stages of rehabilitation when pain or pathology might preclude high load exercises and thus gradually reduces the symptoms.
  Other Names: Sphymomanometer
  Arms: DNF Group
Procedure: Muscle Energy Technique — MET was applied to Upper trapezius, Levator scapulae and Scalene Following the 7-10 seconds isometric contraction and complete relaxation of all elements, the stretch is maintained for 30 seconds. The effort and the counter-pressure should be modest (20% of available strength) and painless. The process is repeated 3-5 times.
  Arms: MET Group
Procedure: Static stretching and Cervical non thrust manipulation — conventional treatment for 5 days per week for 2 weeks such as MHP (Moist Heat Pack) for 20 minutes, Static Stretching exercises for upper trapezius, levator scapulae and scalene muscle which is held for 10-30 seconds- repeated 3-5 times, Cervical spine non-thrust mobilization (Grade 3) was given to each segment from C2-C7 was oscillated for 10 repetitions, followed by a 10 seconds rest between segments, Cervical spine active ROM (Range of Motion) exercises with 10 repetitions- 2-3 times a day and Postural exercises were given as home programme.
  Arms: Conventional group

SUMMARY:
A long term habitual posture with abnormal loading of ligaments and muscles, leads to development of neck pain. 33 patients including 18 males and 15 females were selected and randomly allocated into three groups using sealed opaque envelope containing treatment allocation. Group A (n=11) received conventional treatment such as MHP (Moist Heat Pack), Static Stretching exercises, Cervical spine non-thrust mobilization, Cervical spine active ROM (Range of Motion) exercises and Postural exercises. Group B (n=11) received DNF training with conventional treatment. Group C (n=11) received Muscle Energy Technique (MET) in additional to conventional treatment. Primary outcome measure functional disabilities and secondary measure pain and ROM were recorded at baseline, 7th day and 14th day.One-way ANOVA was used for within group analysis. Repeated measure ANOVA followed by post hoc analysis was employed for between group comparisons. The results suggest that there was a significant improvement in mean change scores of Neck Disability Index (NDI), Visual Analogue Scale (VAS) and Range of Motion (ROM) .Both DNF training and MET have additional therapeutic effects over a standard care by reducing functional disabilities, pain and in improving ROM in mechanical neck pain patients.

DETAILED DESCRIPTION:
According to Janda, postural muscles have tendency to get shorten, in both normal and pathological conditions. Upper trapezius, levator scalpulae and scalene are most common postural muscles. Additionally, longus colli and longus capitis (DNF) have important role in postural support and their impaired activation leads to neck pain.

More recently, muscle based treatments approaches for MNP evolved from a passive treatment technique such as myofascial release towards more active treatment technique such as MET and DNF training.

Group A (N=11) received conventional treatment for 5 days per week for 2 weeks such as MHP (Moist Heat Pack) for 20 minutes, Static Stretching exercises for upper trapezius, levator scapulae and scalene muscle which is held for 10-30 seconds- repeated 3-5 times, Cervical spine non-thrust mobilization (Grade 3) was given to each segment from C2-C7 was oscillated for 10 repetitions, followed by a 10 seconds rest between segments, Cervical spine active ROM (Range of Motion) exercises with 10 repetitions- 2-3 times a day and Postural exercises were given as home programme.

Group B (N=11) received DNF training along with conventional treatment. In this programme, emphasis was placed on first attaining the correct craniocervical flexion action, with minimal activity of the superficial cervical flexor muscles. The craniocervical flexion action involves a specific craniocervical movement (nodding - "yes" movement) of head such that it remains in contact with the supporting surface. Once the correct action had been achieved, participants were instructed in the use of the sphygmomanometer to guide the training of the Craniocervical Flexors muscle contraction at the various incremental levels of pressure (22 to 30 mmHg, progressively inner range positions).

Group C (N=11) received MET in additional to conventional treatment. MET was applied to Upper trapezius, Levator scapulae and Scalene Following the 7-10 seconds isometric contraction and complete relaxation of all elements, the stretch is maintained for 30 seconds. The effort and the counter-pressure should be modest (20% of available strength) and painless. The process is repeated 3-5 times.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years
* Neck pain of minimum duration of six weeks
* Both males and females
* Signed informed consent form
* Tightness of upper trapezius, levator scapulae, scalene muscles on painful side
* Should not be recieving any other therapeutic intervention
* Should not be on medication
* Willing to participate

Exclusion Criteria:

* Inflammatory, Malignant and Neurological conditions
* Metabolic disease
* Neck pain radiating into arms and upper extremity
* Neck pain associated with headaches or facial pain
* Recent major trauma or fracture of the cervical spine
* Referred pain
* History of surgery of cervical spine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Functional disabilities (Neck Disability Index (NDI) | 2 Weeks
  Neck Disability Index (NDI):
  It is a self reported ten-item scale. Each item assess different neck pain complaints. Most of the items are related to restrictions in activities of daily living, and each item is expressed by 6 different assertions in the range 0-5, with 0 indicating no disability and 5 indicating highest disability. The total score ranges from 0 to 50. The scale was measured at baseline, 7th day and 14th day.

SECONDARY OUTCOMES:
Pain (Visual Analogue Scale (VAS) | 2 Weeks
  Visual Analogue Scale (VAS):
  It was use assess the severity of pain. A 10 cm horizontal line was drawn, with 0 means no pain and 10 means the worst possible pain. The patient was asked to mark a point the scale representing their intensity of pain. The scale was measured at baseline, 7th day and 14th day.
Range of Motion (ROM) | 2 Weeks
  Goniometric measurement:
  Active range of motion was assessd using universal standard goniometer for cervical flexion, extension, side flexion (left and right), rotation (left and right). All ranges were assessed in sitting position and the data was collected at baseline, 7th day and 14th day.

CONTACTS AND LOCATIONS:
Overall Officials: Harshita Yadav, M.P.T, Principal Investigator — Maharishi Markandeshwar University, Mullana-Ambala
Locations (1):
- Harshita Yadav, Ambāla, Haryana, India